CLINICAL TRIAL: NCT03143257
Title: Ambispective Clinical Evaluation of Sophono™
Acronym: ACES
Status: Completed | Type: Observational
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16043ENT
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Conductive Hearing Loss; Single-Sided Deafness; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects: Diagnosed with Conductive Hearing Loss (CHL), Single-Sided Deafness (SSD)and mixed Hearing Loss (HL) who currently have or have had the Sophono implant
  Interventions: Device: Sophono Bone Conduction Hearing Systems

INTERVENTIONS:
Device: Sophono Bone Conduction Hearing Systems — The Sophono Bone Conduction Hearing Systems are a family of sound processors and accessories that operate on the principle of Bone Conduction (BC) of sound vibrations. The Sophono Bone Conduction Hearing Systems transmits audio vibrations through the skin into the bone where sound is sensed by the inner ear/cochlea.
  The Sophono Sound Processor is magnetically attracted to the Magnetic Implant and Magnetic Spacer. The Magnetic Implant, which is secured to the skull bone, affixes the Magnetic Spacer to the head transcutaneously through magnetic attraction forces, and the Sound Processor is magnetically affixed to the Magnetic Spacer. Vibration from the Sound Processor is transduced through the Magnetic Spacer to the Magnetic Implant and through the bone to the inner ear.

SUMMARY:
Study to accumulate post-market clinical evidence for the safety and effectiveness of the Sophono Alpha 2 and Alpha 2 Maximum Power Output (MPO) systems in subjects diagnosed with conductive hearing loss, single-sided deafness and mixed hearing loss who currently have or have had the Sophono implant.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who currently has or who has had the Sophono implant (including those who have been explanted)
* Has or has had Sophono implant for 3 months or longer

Exclusion Criteria:

* Subject has implant but is unable or unwilling to perform audiologic testing
* Subject is currently participating in another clinical study and has not been approved for concurrent enrollment by the Study Sponsor

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The subject population for this study includes male and female patients 5 years of age and older who have received the Sophono implant. Subjects will be recruited from Investigators who have implanted Sophono systems or from other non-investigator physician referrals. Subjects are expected to represent a population diagnosed with conductive hearing loss (CHL), single-sided deafness (SSD), and mixed hearing loss (HL).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Macias Otology, Phoenix, Arizona
  - UF Health ENT and Allergy, Gainesville, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Park Avenue Otology/Neurotology, New York, New York
  - Carolina Ear & Hearing Clinic, Raleigh, North Carolina
  - Pittsburgh Ear Associates, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sophono Implant: All Study Participants that have had a previous Sophono Bone Conduction Hearing System implant. No interventions were administered.
Period: Overall Study
Arm/Group | Sophono Implant
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 71 participants were enrolled, 3 presented with bilateral device use which amounted to 74 enrolled ears.
Units Other Than Participants: Ears
Groups:
- All Participants: All Study Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Number analyzed (Ears) | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23.1 [9 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome Measure: Proportion of Adverse Events (AEs) Related to Sophono Implant
Description: The primary safety endpoint is the proportion of AEs related to the Sophono implant, which will be assessed through retrospective surgical chart review and prospective Ear, Nose and Throat (ENT) exam.
Time Frame: From Implantation to Study Visit, up to 6 years
Measure: Number (95% Confidence Interval); unit: Proportion of Adverse Events
Arm/Group | All Participants
Number analyzed (Participants) | 71
Proportion of Adverse Events | 0.038 [0.018 to 0.070]

2. Primary Outcome: Gain in Sensitivity to Sound in Decibels (dB) Resulting From Sophono Alpha 2 Maximum Power Output (MPO) Processor
Description: The primary efficacy endpoint is the difference (gain) in the free-field pure tone audiometry assessed by pure tone average (PTA) unaided (AC) and aided (BC) by the Alpha 2 MPO processor. Standard audiometry test was used to assess free field pure tone audiometry.
Time Frame: 1 day
Population: 69 participants had prospective data (72 ears) and no data was obtained for 2 subjects (deviations noted) so the number of ears analyzed was 70 (67 subjects).
Measure: Mean (Standard Deviation); unit: decibles
Units Other Than Participants: Ears
Groups:
- None AC: Unaided without the processor (Air Conduction)
- None BC: Unaided without the processor (Bone Conduction)
- Aided Alpha 2: Aided Alpha 2
- Aided Alpha 2 MPO: Aided Alpha 2 MPO Processor
Arm/Group | None AC | None BC | Aided Alpha 2 | Aided Alpha 2 MPO
Number analyzed (Participants) | 67 | 67 | 67 | 67
Number analyzed (Ears) | 70 | 70 | 70 | 70
decibles | 79.1 (21.4) | 41.2 (26.8) | 39.4 (11.2) | 35.7 (11.0)
Statistical Analysis 1: Comparison: None AC vs None BC; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 38.0, Standard Deviation 16.1
Statistical Analysis 2: Comparison: None AC vs Aided Alpha 2 MPO; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 43.5, Standard Deviation 20.0
Statistical Analysis 3: Comparison: Aided Alpha 2 vs Aided Alpha 2 MPO; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 3.7, Standard Deviation 5.0

3. Secondary Outcome: Compare the Effectiveness of the Sophono Alpha 2 Processor to the Alpha 2 MPO Processor
Description: All participants were tested with both the Alpha 2 and Alpha 2 MPO processor and also with no processor (Air Conduction) and a standard lab vibration device (Bone Conduction). The difference in the free-field pure tone audiometry assessed by PTA aided by Alpha 2 processor compared to the PTA aided by Alpha 2 MPO processor.
Time Frame: 1 day
Population: 69 subjects (N=72 implanted ears) were used to evaluate the primary effectiveness endpoint. 69 of 71 enrolled subjects were included in the effectiveness analysis. Two subjects did not have prospective data available: one did not have prospective audiologic exams completed and the other subject had audiologic data removed from analysis at the recommendation of the treating sub-investigator who felt the data collected to be inaccurate based on subject response.
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: ears
Groups:
- No Processor (Air Conduction); Standard Vibration Device (Bone Conduction); Alpha 2 Processor; Alpha 2 MPO Processor: The processors were tested in random order (e.g. subjects were tested with both the Alpha 2 processor and the Alpha 2 MPO processor separately but in random order). The participant was unaware which was being used for each test (the processors look the same, differences are internal and not visible). The tests were conducted four times, once for each processor and once with no processor (Air Conduction) and once with the lab standard vibration device (Bone Conduction).
Arm/Group | No Processor (Air Conduction) | Standard Vibration Device (Bone Conduction) | Alpha 2 Processor | Alpha 2 MPO Processor
Number analyzed (Participants) | 69 | 69 | 69 | 69
Number analyzed (ears) | 72 | 70 | 70 | 70
dB | 70.9 (16.7) | 33.5 (23.2) | 39.5 (11.1) | 36.0 (11.1)

4. Secondary Outcome: Percentage of Participants Satisfied After System Use
Description: Subject satisfaction, via non-validated satisfaction questions
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 68
percentage of participants
  Satisfied with the processor | 63
  Satisfied with appearance | 74
  Would recommend device to another patient | 79

5. Secondary Outcome: Assess QOL After System Use
Description: QOL assessment through validated Abbreviated Profile of Hearing Aid Benefit (APHAB)™ assessment. The APHAB is a questionnaire with four subscales (Ease of Communication, Reverberation, Background Noise, and Aversiveness). Items are answered on a seven-point scale from "always" to "never". Scores for subscales can range from 0% (no difficulty) to 99% (maximum difficulty). Negative scores reflect a better benefit from aided hearing all subcategories are reported in percentiles. Abbreviated Profile of Hearing Aid Benefit was taken at 1 time point. Per request of site Institutional Review Board (IRB) pediatric patients were given a pediatric version. Calculation compared aided to unaided hearing.
  A global score is computed by averaging the East of Communication, Reverberation, and Background Noise scale scores. Questions are answered for unaided and aided listening. Aided scores are subtracted from unaided scores.
Time Frame: 1 day
Population: In this study 63 of 71 subjects completed the APHAB.
Measure: Mean (Standard Deviation); unit: Percentage of Score (hearing problem)
Units Other Than Participants: Subject Responses
Groups:
- Aided With Processor: In this arm all participants responded to the questions based on when they are wearing their own Sophono device (i.e. either the Sophono Alpha 2 or the Alpha 2 MPO).
- Unaided Without Processor: In this arm all participants responded to the questions based on when they are not wearing their own hearing device.
Arm/Group | Aided With Processor | Unaided Without Processor
Number analyzed (Participants) | 63 | 63
Number analyzed (Subject Responses) | 63 | 63
Percentage of Score (hearing problem)
  Ease of Communication (%) | 25.4 (21.7) | 49.1 (28.3)
  Reverberation (%) | 32.4 (17.2) | 53.7 (19.8)
  Background Noise (%) | 33.0 (20.3) | 63.6 (20.5)
  Aversiveness (%) | 44.3 (25.6) | 31.5 (23.7)
  Global Score (%) | 30.3 (16.3) | 55.3 (20.1)
Statistical Analysis 1: Comparison: Aided With Processor vs Unaided Without Processor; Test type: Superiority; Overall Benefit Score = -15, Standard Deviation 18.5 — The overall benefit can be determined by subtracting the aided and unaided scores of Ease of Communication, Reverberation, Background Noise & Aversiveness. A negative score in overall benefit indicates a positive benefit to the subject

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from each subject at the single study visit which occurred at a range of 3 months to 5 years post-implantation. The collective Adverse Events in this study represent a range of time from implantation to the study visit (3 months to 5 years post implantation).
Description: All adverse events present at the prospective visit were collected. Only treatment (surgical procedure or device) related events were collected retrospectively.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 9/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=71)
Implant Site Pain (Skin and subcutaneous tissue disorders) | 2
Incision Site Erythema (Skin and subcutaneous tissue disorders) | 1
Medical Device Site Discomfort (Skin and subcutaneous tissue disorders) | 4
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03143257/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03143257/SAP_001.pdf